CLINICAL TRIAL: NCT00971867
Title: Rollover Study of Weekly Paclitaxel (BMS-181339) in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-539
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Solution, I.V., 100 mg/m2 Weekly for 6 of 7 weeks, Until disease progression or unacceptable toxicity became apparent
  Other Names: Taxol; BMS-181339

SUMMARY:
The purpose of this study is to provide access to paclitaxel therapy to subjects with advanced head and neck cancer who have completed the previous late phase 2 study (CA139-388) and should have continued therapy with paclitaxel as the discretion of the investigator, and to evaluate the frequency and the severity of observed adverse reactions in treated subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced head and neck cancer who have completed the previous late phase 2 study (CA139-388) and should have continued therapy with paclitaxel as the discretion of the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-08-04 (Actual); Primary Completion 2008-11-26 (Actual); Study Completion 2008-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- Japan (9):
  - Local Institution, Kashiwa-shi, Chiba
  - Local Institution, Matsuyama, Ehime
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Osaka, Osaka
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Meguro-ku, Tokyo
  - Local Institution, Kanagawa
  - Local Institution, Tochigi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 Participants Treated
Groups:
- Paclitaxel: Each vial (16.7 mL) contains 100 mg
Period: Overall Study
Arm/Group | Paclitaxel
Started | 11
Completed | 0
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Participant Withdrew Consent | 1
Not completed — Disease Progression | 6

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With SAEs
Description: Number of Participants with SAEs
Time Frame: From the first infusion to the completion of study. Approximately up to 28 months
Population: All Treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Number of Participants | 3

2. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: Number of Participants with Adverse Events Leading to Discontinuation
Time Frame: From the first infusion to the completion of study. Approximately up to 28 months
Population: All Treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Number of Participants | 5

3. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: From the first infusion to the completion of study. Approximately up to 28 months
Population: All Treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Number of Participants | 11

4. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Number of Participants with Laboratory Abnormalities
Time Frame: From the first infusion to the completion of study. Approximately up to 28 months
Population: All Treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Number of Participants | 11

5. Primary Outcome: Number of Participants With Drug Related Laboratory Abnormalities
Description: Number of Participants with Drug Related Laboratory Abnormalities
Time Frame: From the first infusion to the completion of study. Approximately up to 28 months
Population: All Treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Number of Participants | 11

6. Secondary Outcome: Number of Participants With Best Overall Response Per RECIST Criteria
Description: Best overall response is represented by the number participants who have had complete response, partial response and have stable disease.
Time Frame: From the enrollment in CA139-388 (NCT00855764) study up to 904 days after the first infusion in CA139-388 study. Approximately up to 42 Months
Population: All Treated Participants in CA139-388 (NCT00855764) and who rolled over into CA139-539
Measure: Number; unit: Number of Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Number of Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 6
  Stable Disease (SD) | 4

7. Secondary Outcome: Number of Participants With Best Overall Response Per the General Rules for Clinical and Pathological Studies of Head and Neck Cancer
Description: Best overall response is represented by the number participants who have had complete response, partial response and not completed.
Time Frame: as for outcome 6
Population: All Treated Participants in CA139-388 (NCT00855764) and who rolled over into CA139-539
Measure: Number; unit: Number of Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Number of Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 9
  Not Completed | 1

8. Secondary Outcome: Duration of Overall Response as Per RECIST Criteria
Description: DOR is defined as the median time from the first date of Partial Response to the first date of Progressive Disease. Participants were evaluated for DOR in a separate study (NCT00971867).
Time Frame: as for outcome 6
Population: All Treated Participants in CA139-388 (NCT00855764) and who rolled over into CA139-539
Measure: Median (Full Range); unit: Days
Arm/Group | Paclitaxel
Number analyzed (Participants) | 11
Days | 222 [70 to 847]

9. Secondary Outcome: Duration of Overall Response as Per the General Rules for Clinical and Pathological Studies of Head and Neck Cancer
Description: as for outcome 7
Time Frame: as for outcome 6
Population: All Treated Participants in CA139-388 (NCT00855764) and who rolled over into CA139-539
Measure: Median (Full Range); unit: Days
Arm/Group | Paclitaxel
Number analyzed (Participants) | 10
Days | 269 [140 to 904]

ADVERSE EVENTS:
Time Frame: From the first infusion to the completion of study. Approximately up to 28 months
Arm/Group | Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=11)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cancer Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=11)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11)
Hypoesthesia (Nervous system disorders) | 9
Fatigue (General disorders) | 7
Weight Disorder (General disorders) | 5
Nail Disorder (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less